CLINICAL TRIAL: NCT05700461
Title: Pilot Study of an Implantable Microdevice for in Situ Evaluation of Drug Response in Renal Cell Carcinoma
Brief Title: Drug Screening Using Novel IMD in Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wenxin Xu (Other)
Responsible Party: Sponsor-Investigator, Wenxin Xu, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-492
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Kidney Cancer
Keywords: Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Kidney Cancer; Suspected Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Implantable microdevice (IMD) + Biopsy + Standard of Care Treatment (Experimental): Participants with confirmed or suspected metastatic Renal Cell Carcinoma (RCC) and who are candidates for standard of care metastatectomy or debulking/consolidative nephrectomy will be selected for study participation and will undergo study procedures as outlined:
  * Placement of 1-6 microdevice(s) 72 +/- 24 hours prior to scheduled, standard of care surgery. The number of microdevices implanted into a tumor will be made on a case-by-case basis based on tumor and participant factors before and during the procedure.
  * At the time of standard of care surgery, surgical removal of microdevice(s) along with surrounding tumor tissue.
  * Monitoring for safety endpoints during inpatient stay and at a follow-up clinic visit.
  Interventions: Combination Product: Implantable Microdevice (IMD)

INTERVENTIONS:
Combination Product: Implantable Microdevice (IMD) — Small, implantable device with 20 microreservoirs for drug and drug combinations, via needle, percutaneously, and guided by interventional radiologic techniques.
  Drugs include all or a subset of the following: Cabozantinib, Pazopanib, Lenvatinib, Axitinib, Ipilimumab, Nivolumab, Pembrolizumab, Carboplatin, Paclitaxel, Abemaciclib, Gemcitabine, Everolimus, Belzutifan, Cabozantinib + nivolumab, Cabozantinib + belzutifan, Ipilimumab + nivolumab, Lenvatinib + pembrolizumab, Lenvatinib + everolimus, Abemaciclib + belzutifan, and Tivozanib.

SUMMARY:
This research is being done to study the safety and feasibility of implanting and retrieving a microdevice that releases microdoses of 19 specific drugs or drug combinations as a possible tool to evaluate the effectiveness of several cancer drugs against metastatic renal cell carcinoma (RCC).

The name of the intervention(s) involved in this study are:

* Implantable Microdevice (IMD)
* Surgery (excision of tumor)
* Drugs used in this study will only include drugs already used as standard of care for the treatment of metastatic renal cell carcinoma (RCC)

DETAILED DESCRIPTION:
This Pilot research is being done to study the safety and feasibility of implanting and retrieving a microdevice that releases microdoses of 19 specific drugs or drug combinations as a possible tool to evaluate the effectiveness of several cancer drugs against metastatic renal cell carcinoma (RCC). The drugs participants receive will include medications currently used as standard-of-care treatment for metastatic RCC as well as medications currently approved in other cancer types that are under investigation for treatment of RCC.

* This study involves planting 1 to 6 microdevices, each small enough to fit inside the tip of a needle, into a tumor. The microdevices will release microdoses of cancer drugs via passive diffusion. The drugs will only penetrate the local tumor tissues.
* After approximately 3 days, the microdevices and small regions of surrounding tissues will be removed and analyzed.

The research study procedures include screening for eligibility, study imaging and evaluations, blood collections, tumor biopsies, and follow up visits.

The U.S. Food and Drug Administration (FDA) has not approved the microdevice as a treatment for any disease.

The drugs being used have been FDA-approved for the treatment of cancers.

Participation in this research study is expected to last up to 4 months.

It is expected that about 5 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have the ability to understand and the willingness to sign a written informed consent document.
* Participants must have confirmed or suspected metastatic renal cell carcinoma, and must be planned for either nephrectomy or metastatectomy as part of their clinical care. The lesion planned for excision must be at least 1cm in size.
* Participants must be 18 years of age or older.
* Participants must be evaluated by a medical oncologist who will determine the clinically appropriate treatment strategy based on clinical history and extent of disease.
* Patients must be deemed medically stable to undergo both percutaneous procedures and standard-of-care surgical procedures.
* Participants will undergo laboratory testing within 30 days prior to the procedure (or within 72 hours if there has been a change in the clinical status since the initial blood draw). Patients must have absolute neutrophil count ≥1,000/mcL, platelets ≥50,000/mcL, PT (INR) 1.5 and PTT <1.5x control.
* Participants must have undergone CT or MRI that assesses the extent of disease and allows the research team to assess for study eligibility. This will have been done as part of the standard-of-care.
* The participant's case must be reviewed by representatives of interventional radiology and the appropriate surgical subspecialty to assess the following factors:

  * Patient is clinically stable to undergo microdevice implantation and surgical procedures
  * Patient has sufficient volume of disease to allow implantation of the microdevice
  * Patient has a lesion for which the microdevice is a) amenable to percutaneous placement, and b) amenable to removal at the time of surgery
* Patients must be willing to undergo research-related genetic sequencing (somatic and germline) and data management, including the deposition of de-identified genetic sequencing data in NIH central data repositories.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, or psychiatric illness/social situations that would limit the safety of a biopsy and/or surgery.
* Uncorrectable bleeding or coagulation disorder known to cause increased risk with surgical or biopsy procedures (detailed below).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Safe Microdevice Procedure | Up to 45 days
  Defined by any grade 3-5 adverse event (AE) associated with microdevice placement or retrieval (attribution possible or higher) based on CTCAEv5.
Number of Patients with Feasible Microdevice Procedure | 72 hours
  Defined as technical success of microdevice placement and microdevice retrieval from the surgery specimen plus having sufficient amount and quality of tissue for histopathology analysis and interpretation of at least 50% of the microdevice reservoirs.

CONTACTS AND LOCATIONS:
Overall Officials: Wenxin Xu, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation.